CLINICAL TRIAL: NCT06415084
Title: Hyperemesis Gravidarum Prevalence : A Repeated Cross-sectional Population Based Study
Brief Title: Prevalence of Hyperemesis Gravidarum
Acronym: PHyperEG1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Effik (Industry); Université d'Auvergne (Other); AUDIPOG (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 VENDITTELLI
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Nausea and Vomiting
Keywords: Nausea vomiting; Pregnancy; Disease prevalence; Hyperemesis gravidarum
MeSH Terms: conditions — Nausea; Vomiting; Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Nausea and vomiting during pregnancy represent one of the most common symptoms of pregnancy, affecting 35 to 91% of women. Most often, the symptoms are mild, without impairment of quality of life and disappear at the end of the first trimester. More severe forms constitute hyperemesis gravidarum (HG) (hyperemesis gravidarum). In approximately 35% of women, nausea and vomiting during pregnancy are disabling, alter daily life and professional activity and negatively affect family relationships. For 0.3 to 3.6% of pregnancies, this vomiting is uncontrollable and constitutes the main cause of hospitalization in the first trimester of pregnancy.

Faced with the incomprehension and lack of knowledge of their illness, both in society and in the medical community, patient associations have been created in France to gain recognition for HG and raise awareness among caregivers and women about this illness and its consequences. Vomiting repeatedly for weeks, losing weight sometimes significantly, being weakened, no longer able to cope with daily life, family life and work, is what some women can experience while they are pregnant and that society tells them : "pregnancy is not an illness".

Although HG is common, its real prevalence is unknown, particularly in France, because there have been few studies involving small samples. A population study is desirable because it is likely that the prevalence of these pregnancy aches differs depending on the country. This subject is important because vomiting during pregnancy has an impact on women's quality of life and their desire to become pregnant again.

The main objective of this observation study is to evaluate the prevalence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum), in the general population, in the first trimester of pregnancy.

The secondary objectives are:

* to assess the prevalence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum), in the second and third trimesters of pregnancy,
* to assess the prevalence of uncomplicated pregnancy-related nausea and/or vomiting in the three trimesters of pregnancy,
* to evaluate the prevalence of hyperemesis gravidarum (with or without hospitalization) in the three trimesters of pregnancy,
* to evaluate the prevalence of hyperemesis gravidarum requiring hospitalization in the three trimesters of pregnancy,
* to evaluate the distribution of nausea and/or vomiting (mild, moderate and severe) according to the modified-PUQE score, in the three trimesters of pregnancy,
* to evaluate the predictive factors for the occurrence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum) in the first trimester of pregnancy,
* to assess health-related quality of life in the event of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum), in the three trimesters of pregnancy,
* and to compare health-related quality of life between women with pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum) and those without, in the first trimester of pregnancy.

DETAILED DESCRIPTION:
Study design: A repeated population based cross sectional survey.

A woman can withdraw from the study early for the following reasons:

* the woman's decision,
* a major protocol deviation,
* and loss to follow-up (a subject lost to follow-up is a participant who did not answer to all the surveys)

The study may be stopped temporarily or permanently for the following reasons:

* Recruitment too low or nonexistent,
* Decision of the sponsor and of the investigator-coordinator.

Methods of recruitment :

The inclusion of women will take place after one of the 1st trimester ultrasounds. They will have to complete, from their home, an online self-questionnaire including, among other things, the modified-PUQE score assessing the severity of nausea and vomiting during the first trimester of pregnancy. Women who have had an early ultrasound, before 10 weeks of amenorrhea (WA), will be re-interviewed at the start of the 2nd trimester via an online questionnaire.

Subsequently, women who responded in the 1st trimester and who present with hyperemesis gravidarum or uncomplicated pregnancy-related nausea and/or vomiting will be questioned, again, about the existence of nausea and vomiting just after the deadline for the 2nd trimester ultrasounds (between 20 WA+0 day and 25 WA+0 day) and 3rd trimester (between 30 WA+0 day and 35 WA+0 day), via an online self-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women having a monitored pregnancy in Auvergne,
* Major,
* Speaking French,
* Socially insured,
* Having given their agreement to participate in the study.

Exclusion Criteria:

* Women refusing to participate in the study,
* Not speaking French,
* Major incapacitated persons.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women are included in this study.
Study Population: Women will be recruited for the study during their first-trimester ultrasound. They will be informed of the study by the sonographer, who will give them the link to access the first online study questionnaire. This questionnaire will enable tthe collect of the women's consent to particpate to the study, after online verification of eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 604 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum) | First trimester of pregnancy (up to 13 weeks of gestation)
  Prevalence of uncomplicated nausea and/or vomiting or with hyperemesis gravidarum. Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6. Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.

SECONDARY OUTCOMES:
Prevalence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum) | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  Prevalence of uncomplicated nausea and/or vomiting or with hyperemesis gravidarum. Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6. Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.
Prevalence of pregnancy-related nausea and/or vomiting (uncomplicated or with hyperemesis gravidarum) | Third trimester of pregnancy (>= 28 weeks of gestation)
  Prevalence of uncomplicated nausea and/or vomiting or with hyperemesis gravidarum. Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6. Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.
Prevalence of uncomplicated pregnancy-related nausea and vomiting | First trimester of pregnancy (up to 13 weeks of gestation)
  Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6.
Prevalence of uncomplicated pregnancy-related nausea and vomiting | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6.
Prevalence of uncomplicated pregnancy-related nausea and vomiting | Third trimester of pregnancy (>= 28 weeks of gestation)
  Uncomplicated pregnancy-related nausea and vomiting is defined as pregnancy-related nausea and vomiting associated with: weight loss < 5%; without clinical signs of dehydration and; a modified-PUQE score ≤ 6.
Prevalence of hyperemesis gravidarum, with or without hospitalization | First trimester of pregnancy (up to 13 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.
Prevalence of hyperemesis gravidarum, with or without hospitalization | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.
Prevalence of hyperemesis gravidarum, with or without hospitalization | Third trimester of pregnancy (>= 28 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7.
Prevalence of hyperemesis gravidarum with hospitalization | First trimester of pregnancy (up to 13 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7. The women are hospitalized.
Prevalence of hyperemesis gravidarum with hospitalization | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7. The women are hospitalized.
Prevalence of hyperemesis gravidarum with hospitalization | Third trimester of pregnancy (>= 28 weeks of gestation)
  Hyperemesis gravidarum is defined as pregnancy-related nausea and vomiting associated with at least one of the following signs: weight loss ≥ 5%; one or more clinical signs of dehydration; a modified-PUQE score ≥ 7. The women are hospitalized.
Distribution of mild, moderate and severe nausea and vomiting | First trimester of pregnancy (up to 13 weeks of gestation)
  Distribution of nausea and vomiting according to the modified-PUQE score: mild (modified-PUQE score ≤ 6), moderate (modified-PUQE score ≥ 7 and ≤ 12) and severe (modified-PUQE score ≥ 13) vomiting.
Distribution of the modified-PUQE score | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  Distribution of nausea and vomiting according to the modified-PUQE score: mild (modified-PUQE score ≤ 6), moderate (modified-PUQE score ≥ 7 and ≤ 12) and severe (modified-PUQE score ≥ 13) vomiting.
Distribution of mild, moderate and severe nausea and vomiting | Third trimester of pregnancy (>= 28 weeks of gestation)
  Distribution of nausea and vomiting according to the modified-PUQE score: mild (modified-PUQE score ≤ 6), moderate (modified-PUQE score ≥ 7 and ≤ 12) and severe (modified-PUQE score ≥ 13) vomiting.
Self-administered "Health-Related Quality of Life for Nausea and Vomiting of Pregnancy" (NVP-QOL) questionnaire | First trimester of pregnancy (up to 13 weeks of gestation)
  The NVP-QOL questionnaire measures health-related quality of life in the last week and contains 30 items covering 4 general domains: physical symptoms and/or aggravating factors (9 items), fatigue (4 items), emotions (7 items), and limitations (10 items). Each item is measured using a 7-point Likert scale from 1 ("none of the time") to 7 ("all the time"). A total score is obtained by summing the scores of each of the 30 items (with reversed score for item 20), and ranges between 30 (corresponding to good QOL) and 210 (corresponding to poor QOL).
Self-administered "Health-Related Quality of Life for Nausea and Vomiting of Pregnancy" (NVP-QOL) questionnaire | Second trimester of pregnancy (between 14 an 27 weeks of gestation)
  The NVP-QOL questionnaire measures health-related quality of life in the last week and contains 30 items covering 4 general domains: physical symptoms and/or aggravating factors (9 items), fatigue (4 items), emotions (7 items), and limitations (10 items). Each item is measured using a 7-point Likert scale from 1 ("none of the time") to 7 ("all the time"). A total score is obtained by summing the scores of each of the 30 items (with reversed score for item 20), and ranges between 30 (corresponding to good quality of life) and 210 (corresponding to poor quality of life).
Self-administered "Health-Related Quality of Life for Nausea and Vomiting of Pregnancy" (NVP-QOL) questionnaire | Third trimester of pregnancy (>= 28 weeks of gestation)
  The NVP-QOL questionnaire measures health-related quality of life in the last week and contains 30 items covering 4 general domains: physical symptoms and/or aggravating factors (9 items), fatigue (4 items), emotions (7 items), and limitations (10 items). Each item is measured using a 7-point Likert scale from 1 ("none of the time") to 7 ("all the time"). A total score is obtained by summing the scores of each of the 30 items (with reversed score for item 20), and ranges between 30 (corresponding to good quality of life) and 210 (corresponding to poor quality of life).
Self-administered "World Health Organization's Quality of Life-BREF " (WHOQOL-BREF) questionnaire | First trimester of pregnancy (up to 13 weeks of gestation)
  The WHOQOL-BREF questionnaire measures generic health-related quality of life in the last two weeks and includes a subset of 26 items. Information from all 26 items is used to calculate scores of four subscales: Physical health, Psychological health, Social relationships, and Environment. Subscales scores range from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Vendittelli, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Reseau de Santé en Périnatalité d'Auvergne, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gadsby R, Barnie-Adshead AM, Jagger C. A prospective study of nausea and vomiting during pregnancy. Br J Gen Pract. 1993 Jun;43(371):245-8. PMID 8373648
- [Background] Einarson TR, Piwko C, Koren G. Quantifying the global rates of nausea and vomiting of pregnancy: a meta analysis. J Popul Ther Clin Pharmacol. 2013;20(2):e171-83. Epub 2013 Jul 13. PMID 23863575
- [Background] Attard CL, Kohli MA, Coleman S, Bradley C, Hux M, Atanackovic G, Torrance GW. The burden of illness of severe nausea and vomiting of pregnancy in the United States. Am J Obstet Gynecol. 2002 May;186(5 Suppl Understanding):S220-7. doi: 10.1067/mob.2002.122605. PMID 12011890
- [Background] Mazzotta P, Stewart D, Atanackovic G, Koren G, Magee LA. Psychosocial morbidity among women with nausea and vomiting of pregnancy: prevalence and association with anti-emetic therapy. J Psychosom Obstet Gynaecol. 2000 Sep;21(3):129-36. doi: 10.3109/01674820009075620. PMID 11076334
- [Background] Eliakim R, Abulafia O, Sherer DM. Hyperemesis gravidarum: a current review. Am J Perinatol. 2000;17(4):207-18. doi: 10.1055/s-2000-9424. PMID 11041443
- [Background] Heitmann K, Nordeng H, Havnen GC, Solheimsnes A, Holst L. The burden of nausea and vomiting during pregnancy: severe impacts on quality of life, daily life functioning and willingness to become pregnant again - results from a cross-sectional study. BMC Pregnancy Childbirth. 2017 Feb 28;17(1):75. doi: 10.1186/s12884-017-1249-0. PMID 28241811
- [Background] Lacasse A, Rey E, Ferreira E, Morin C, Berard A. Validity of a modified Pregnancy-Unique Quantification of Emesis and Nausea (PUQE) scoring index to assess severity of nausea and vomiting of pregnancy. Am J Obstet Gynecol. 2008 Jan;198(1):71.e1-7. doi: 10.1016/j.ajog.2007.05.051. PMID 18166311
- [Background] Lacasse A, Berard A. Validation of the nausea and vomiting of pregnancy specific health related quality of life questionnaire. Health Qual Life Outcomes. 2008 May 9;6:32. doi: 10.1186/1477-7525-6-32. PMID 18471301
- [Background] Dochez V, Dimet J, David-Gruselle A, Le Thuaut A, Ducarme G. Validation of specific questionnaires to assess nausea and vomiting of pregnancy in a French population. Int J Gynaecol Obstet. 2016 Sep;134(3):294-8. doi: 10.1016/j.ijgo.2016.01.023. Epub 2016 May 19. PMID 27262942
- [Background] Baumann C, Erpelding ML, Regat S, Collin JF, Briancon S. The WHOQOL-BREF questionnaire: French adult population norms for the physical health, psychological health and social relationship dimensions. Rev Epidemiol Sante Publique. 2010 Feb;58(1):33-9. doi: 10.1016/j.respe.2009.10.009. Epub 2010 Jan 21. PMID 20096515